CLINICAL TRIAL: NCT01496534
Title: Phase Ib Study of Dovitinib in Combination With Gemcitabine Plus Cisplatin or Gemcitabine Plus Carboplatin in Patients With Advanced Solid Tumors
Brief Title: Phase Ib Study of Gemcitabine Plus Cisplatin or Carboplatin Plus Dovitinib in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: toxicity of combination of medications
Sponsor: Matthew Galsky (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 11-0946
Record Dates: First submitted 2011-12-12; First posted 2011-12-21 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Solid Tumors; Bladder Cancer
Keywords: advanced solid tumors; bladder cancer; gemcitabine; cisplatin; carboplatin; solid tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisplatin (Active Comparator): Gemcitabine 1000 mg/m2 IV on days 1 + 8 Cisplatin 70 mg/m2 IV day 1 Dovitinib given orally on days 1-5, 8-12 and 15-19. Treatment will be recycled every 21-days. The dose of dovitinib will be escalated in successive cohorts.
  Interventions: Drug: Cisplatin
- Carboplatin (Active Comparator): Gemcitabine 1000 mg/m2 IV on days 1 + 8 Carboplatin AUC 5 IV day 1 Dovitinib given orally on days 1-5, 8-12 and 15-19. Treatment will be recycled every 21-days. The dose of dovitinib will be escalated in successive cohorts.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Cisplatin — Gemcitabine 1000 mg/m2 IV on days 1 + 8 Cisplatin 70 mg/m2 IV day 1 Dovitinib given orally on days 1-5, 8-12 and 15-19. Treatment will be recycled every 21-days. The dose of dovitinib will be escalated in successive cohorts
  Other Names: TKI258
  Arms: Cisplatin
Drug: Carboplatin — Gemcitabine 1000 mg/m2 IV on days 1 + 8 Carboplatin AUC 5 IV day 1 Dovitinib given orally on days 1-5, 8-12 and 15-19. Treatment will be recycled every 21-days. The dose of dovitinib will be escalated in successive cohorts
  Other Names: TKI258
  Arms: Carboplatin

SUMMARY:
This is a phase Ib dose escalation study of dovitinib given in combination with either gemcitabine plus cisplatin or carboplatin in patients with advanced solid tumors. Patients with advanced solid tumors, for whom treatment with gemcitabine plus cisplatin or carboplatin would otherwise be warranted, will be enrolled. The dose of dovitinib will be escalated in successive cohorts using standard "3+3" dose escalation rules. Patients will continue treatment, in the absence of prohibitive toxicity, until disease progression. The study will define the recommended phase II dose of these combination regimens.

DETAILED DESCRIPTION:
This is a phase Ib study of dovitinib given in combination with gemcitabine plus cisplatin or carboplatin in patients with advanced solid tumors. This study will utilize standard 3+3 dose escalation rules to define the recommended phase II dose. Dose escalation will proceed independently in the two cohorts (cisplatin cohort: gemcitabine + cisplatin + dovitinib; carboplatin cohort: gemcitabine + carboplatin + dovitinib). Patients will receive treatment for up to 6 cycles, in the absence of toxicity, until disease progression

Primary Objective:

To determine the recommended phase II dose of dovitinib given in combination with gemcitabine plus cisplatin or carboplatin.

Secondary Objectives:

* To determine the response rate to treatment as per Response Evaluation Criteria in Solid Tumors (RECIST)
* To determine the toxicity of treatment at per the Common Terminology for Adverse Events (CTCAE v4)
* To determine the pharmacokinetics of dovitinib in combination with gemcitabine plus cisplatin or carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* Karnofsky Performance Status of ≥ 70%.
* Advanced/metastatic solid tumor for which treatment with gemcitabine plus carboplatin or gemcitabine plus cisplatin would otherwise be warranted.
* Prior treatment with chemotherapy is permitted. Patients must not have received more than three prior chemotherapeutic regimens.
* Adequate organ function as determined by the following laboratory values:

  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 100 x 109/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Creatinine of ≤ 1.5 OR Calculated creatinine clearance of ≥ 60 cc/min for the cisplatin cohort.

Calculated creatinine clearance of ≥ 30 cc/min for the carboplatin cohort.

* Bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) ≤ 1.5 ULN
* Alanine Aminotransferase (ALT, SGPT) < 1.5 ULN
* INR ≤ 1.5 and a PTT within normal limits
* LVEF assessed by 2-D echocardiogram (ECHO) > 50% or lower limit of normal or multiple gated acquisition scan (MUGA) > 45% or lower limit of normal

Exclusion Criteria:

* Prior treatment with more than three prior chemotherapy regimens.
* Has had major surgery within 30 days of starting the study treatment
* Have active CNS metastases.
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* Prior cancer treatment must be completed at least 30 days prior to being registered for protocol therapy and the subject must have recovered from the acute toxic effects of the regimen.
* Prior radiation therapy must be completed at least 30 days prior to being registered for protocol therapy.
* Pregnant or breastfeeding.
* Clinically significant infections as judged by the treating investigator.
* Impaired cardiac function or clinically significant cardiac diseases
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patients who are currently receiving anticoagulation treatment with therapeutic doses of warfarin
* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception.
* Fertile males not willing to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of combination regimen | Within the first 21 days of treatment
  The primary objectives of this study are to determine the recommended phase II dose of dovitinib given in combination with gemcitabine plus carboplatin or cisplatin.

SECONDARY OUTCOMES:
Antitumor activity | After every 2 cycles (42 days) of combination therapy up to 3 years
  A CT scan of the chest, abdomen, and pelvis will be performed after every 2 cycles (or sooner if there is evidence of disease progression) while on combination therapy until disease progression (eg, after cycle 2, after cycle 4, and after cycle 6). Response to treatment will be determined using RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Galsky, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Turner N, Grose R. Fibroblast growth factor signalling: from development to cancer. Nat Rev Cancer. 2010 Feb;10(2):116-29. doi: 10.1038/nrc2780. PMID 20094046
- [Background] Knowles MA. Novel therapeutic targets in bladder cancer: mutation and expression of FGF receptors. Future Oncol. 2008 Feb;4(1):71-83. doi: 10.2217/14796694.4.1.71. PMID 18241002
- [Background] Sarker D, Molife R, Evans TR, Hardie M, Marriott C, Butzberger-Zimmerli P, Morrison R, Fox JA, Heise C, Louie S, Aziz N, Garzon F, Michelson G, Judson IR, Jadayel D, Braendle E, de Bono JS. A phase I pharmacokinetic and pharmacodynamic study of TKI258, an oral, multitargeted receptor tyrosine kinase inhibitor in patients with advanced solid tumors. Clin Cancer Res. 2008 Apr 1;14(7):2075-81. doi: 10.1158/1078-0432.CCR-07-1466. PMID 18381947